CLINICAL TRIAL: NCT00656318
Title: Impact of Oral Contraceptives on GABA and Neurosteroids
Status: Terminated | Type: Observational
Why Stopped: Funding withdrawn from study sponsor.
Sponsor: Yale University (Other)
Responsible Party: C. Neill Epperson, M.D., Yale University School of Medicine Department of Psychiatry
Other Study IDs: 0701002178
Record Dates: First submitted 2008-04-07; First posted 2008-04-11 (Estimated); Last update posted 2009-08-25 (Estimated); Status verified 2009-08

CONDITIONS: Healthy
Keywords: women; menses; oral contraceptives; Healthy menstruating females
MeSH Terms: interventions — Contraceptives, Oral; SC-11800 EE; ovcon 35

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Group 1 (Zovia): Subjects will be randomized to receive either the oral contraceptive pill (OCP) Zovia or Necon for 2 months. Prior to beginning the OCP, women will undergo 1 imaging scan. Upon completion of the scan they will receive their first dose of their OCP. Three hours later they will undergo a 2nd imaging scan. Each scan last approximately 1 hour and 15 minutes. This test day is typically scheduled on a Saturday, and lasts approximately 7 hours. Upon completion of the Saturday test day, subjects will remain on their OCP for the remainder of that month and continue taking the pill for a 2nd month. At the end of the 2 months on the pill, subjects will have the option of discontinuing the pill or receiving 1 additional month at no charge before being discharged from the study.
  Interventions: Other: oral contraceptive pill (OCP; OCPs)
- Group 2 (Necon): Subjects will be randomized to receive either the oral contraceptive pill (OCP) Zovia or Necon for 2 months. Prior to beginning the OCP, women will undergo 1 imaging scan. Upon completion of the scan they will receive their first dose of their OCP. Three hours later they will undergo a 2nd imaging scan. Each scan last approximately 1 hour and 15 minutes. This test day is typically scheduled on a Saturday, and lasts approximately 7 hours. Upon completion of the Saturday test day, subjects will remain on their OCP for the remainder of that month and continue taking the pill for a 2nd month. At the end of the 2 months on the pill, subjects will have the option of discontinuing the pill or receiving 1 additional month at no charge before being discharged from the study.
  Interventions: Other: oral contraceptive pill (OCP; OCPs)

INTERVENTIONS:
Other: oral contraceptive pill (OCP; OCPs) — Daily administration of oral contraceptive pill for up to 3 months (2 months of daily administration required for the study).
  Other Names: Zovia 1/35; Necon

SUMMARY:
Thus, the proposed study has the following Specific Aims and Hypotheses:

1. To determine in menstruating women ages 18-45 whether an OCP containing ethinyl estradiol (EE) and the progestin ethinydiol diacetate (ED) increases cortical GABA concentrations as measured using proton magnetic resonance spectroscopy (1H-MRS) above that of an OCP containing EE and the progestin norethindrone (NOR).
2. To determine the relationship between changes in occipital GABA concentrations with acute OCP administration and negative affect with chronic OCP administration over two menstrual cycles.

DETAILED DESCRIPTION:
Approximately 11.6 million women in the United States use oral contraceptives (OCs) each year. The vast majority of OCs combine both estrogen and a type of progestin, or progesterone-like substance into one pill which is taken daily. Depression or a negative change in mood, apparently resulting from the use of OCs, is thought to be one of the main reasons women miss pills or stop taking their oral contraceptive pills (OCPs) altogether. Clinical observation that some women develop depression when taking progestin only OCs or when adding progestins to menopausal estrogen therapy has led to the speculation that the progestin is the likely culprit of these negative mood changes in women using combined OCPs.

The current study is designed to investigate the role of progestins in the development of mood symptoms in OCP users. Women participating in this study will receive one of two different OCPs for three months. Their mood while taking the OCPs will be compared to their mood prior to using OCPs. In addition, each woman will undergo a brain imaging study after the first dose of their OCP to determine whether acute changes in brain chemistry in response to the OCP predicts change in mood with OCP use. By choosing OCPs with the same estrogen product but 2 different types of progestins we hope to determine whether one type of progestin is more likely to result in negative mood.

Determining factors that contribute to the emergence of depression with OC use is the first step in developing newer oral contraceptives that do not have this health outcome and will ultimately improve compliance with OCP use. Reducing side effects of OCPs is likely to improve compliance and thus decrease the prevalence of unwanted pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 - 42 years old and able to give voluntary written informed consent.
* Willing to complete a daily log of mood symptoms for 3 consecutive menstrual cycles.
* Be off of OCPs for at least 3 menstrual periods prior to beginning the study and be willing to go on OCPs for the study.
* Provide documentation of a normal PAP smear, pelvic and breast examination within the previous 12 months prior to enrollment.
* Have regular menstrual cycles 28 to 32 days in length prior to enrollment. The screening cycle must be ovulatory as confirmed by plasma progesterone levels of >3 ng/ml during the luteal phase.
* Negative pregnancy blood test at admission; negative urine pregnancy test on the MRS testing day.

Exclusion Criteria:

* Presence of any DSM-IV Axis I disorder, excepting possible mild to moderate PMS/PMDD, within the previous 12 months.
* Lifetime history of any psychotic disorder, including bipolar disorder.
* Meeting DSM-IV criteria for psychoactive substance (including nicotine) abuse/dependence within the preceding 6 months.
* A history of serious medical or neurological illness, including (but not limited to) major cardiovascular disease, hypertension (SBP > 140 mm Hg and DBP > 90 mm Hg), intracranial mass lesions, seizure disorder, severe hepatic or renal disease, unstable endocrine or metabolic disease, unstable hematologic disease, gynecologic cancer and gallbladder disease, venous thromboembolism, and stroke.
* Diabetes if present with one other cardiovascular risk factor such as hypercholesterolemia or hypertension.
* Hypercholesterolemia if LDL > 160 mg/dl.
* Use of any psychotropic medication within the previous month.
* Alcohol consumption greater than 7 drinks/week.
* Current pregnancy or planning to become pregnant during the course of the study.
* Metallic implants.
* History of or suspected claustrophobias.
* Migraine headaches if > 35 yo.
* Weigh >300 lbs (the 4T magnet has a weight limit <300 lbs)

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women between the ages of 18 and 42 with regular menstrual cycles of 28-32 days will be invited to participate in a brain imaging study examining the effects of two different oral contraceptives on cortical GABA levels.
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2008-08; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
The purpose of this study is to investigate the effect of oral contraceptive pills (OCPs) on cortical GABA concentrations as measured by proton magnetic resonance spectroscopy (1H-MRS) in non-depressed, healthy menstruating women. | Outcomes will be measured at several points during each participants menstrual cycle.

SECONDARY OUTCOMES:
To determine the impact of OCP use on plasma and cerebral spinal fluid (CSF) levels of estradiol (E2) and progesterone, as well as neurosteroids such as pregnenolone, allopregnanolone, pregnanolone and 5 alpha-dihydroprogesterone (5α-DHP). | Outcome will be assessed at several time points for each participant.

CONTACTS AND LOCATIONS:
Overall Officials: C. Neill Epperson, M.D., Principal Investigator — Yale University School of Medicine, Department of Psychiatry
Locations (1):
- Yale University School of Medicine, New Haven, Connecticut, United States